CLINICAL TRIAL: NCT05810376
Title: Effects of Digital-based Physical Activity Intervention on Pain, Function and Exercise Adherence in Individuals With Knee Osteoarthritis: a Randomized Controlled Trial
Brief Title: Effects of Digital-based Physical Activity Intervention in Individuals With Knee Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Hakan Akgul, Mr, Trakya University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021/291
Record Dates: First submitted 2023-03-30; First posted 2023-04-12 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-03

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Patient Education as Topic; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Experimental group will receive patient education, exercise, and digital-based physical activity intervention.
  Interventions: Behavioral: Digital-based physical activity intervention; Other: Patient education and exercise
- Control Group (Active Comparator): Control group will receive patient education and exercise.
  Interventions: Other: Patient education and exercise

INTERVENTIONS:
Behavioral: Digital-based physical activity intervention — The digital behavioral program comprises goal planning, motivational messages and video calls, social support, and routine follow-up of weekly goals.
  Arms: Experimental Group
Other: Patient education and exercise — Patient education will include information on osteoarthritis, prognosis, pain management, importance of physical activity and exercise. The exercise program will include warm up, stretching and strengthening.

SUMMARY:
Physical activity is recommended in the guidelines to improve pain and function in the treatment of knee OA, regardless of the severity of the disease, but still, patients rarely do enough physical activity. The choice of intervention to improve symptoms and disorders may be key to increasing the level of physical activity. Adapting physical activity to the patient's needs and preferences can improve compliance and outcomes. In a Delphi study, the only statement that received 100% support was stated as "Individualized exercise is an integral component of treatment for anyone with osteoarthritis". However, healthcare providers often recommend physical activity programs that do not place too much emphasis on the patient's preferences. The decision to engage in physical activity is multifactorial, and it is necessary to understand people's physical activity preferences better in order to increase participation and compliance.

Digital health interventions have the potential to address physical inactivity as they are accessible to a large part of the population and can be delivered with high efficiency at a low cost. By enabling patient education, support for self-management, motivation, follow-up, feedback and communication, it can prevent, cure or treat many chronic conditions. These features can increase patient motivation and encourage compliance with home exercises and physical activity. Digital behavior change interventions use digital technologies (such as websites, mobile apps, SMS or wearables) to promote and maintain health and have the potential to overcome many barriers compared to in-person programs by providing cost-effective, effective, and accessible information. No study has been found in Turkey examining digital interventions or walking programs that include behavior change techniques to increase physical activity in patients with knee osteoarthritis. Considering environmental, cultural and economic factors in this patient group in our society, we think that walking, which we think is the most appropriate physical activity method in terms of cost, accessibility and equipment, should be a permanent behavior.

Our aim in the study; To examine the effects of digitally assisted physical activity intervention on pain, functionality and exercise commitment in individuals with knee osteoarthritis.

DETAILED DESCRIPTION:
Functional capacity and quality of life decrease in individuals with knee osteoarthritis (OA). This is due to loss of strength and physical inactivity caused by pain or fatigue. Increasing levels of physical activity have been shown to reduce these problems. Another reason why individuals with osteoarthritis have a lower level of physical activity than the general population may be the fear of moving with the thought of more pain. However, physical activity is recommended as a basic treatment for osteoarthritis (Shih, Hootman et al. 2006).

Physical activity is recommended in the guidelines to improve pain and function in the treatment of knee OA, regardless of the severity of the disease, but still, patients rarely do enough physical activity (Zhang, Moskowitz et al.

2008, Zhang, Doherty et al. 2010, Dunlop, Song et al. al. 2011). The choice of intervention to improve symptoms and disorders may be key to increasing the level of physical activity. Adapting physical activity to the patient's needs and preferences can improve compliance and outcomes. In a Delphi study, the only statement that received 100% support was stated as "Individualized exercise is an integral component of treatment for anyone with osteoarthritis" (French, Bennell et al. 2015). However, healthcare providers often recommend physical activity programs that do not place too much emphasis on the patient's preferences. The decision to engage in physical activity is multifactorial, and it is necessary to understand people's physical activity preferences better in order to increase participation and compliance (Holden, Nicholls et al. 2009, Dierckx, Deveugele et al. 2013, Pinto, Danilovich et al. 2017).

Digital health interventions have the potential to address physical inactivity as they are accessible to a large part of the population and can be delivered with high efficiency at a low cost (Iribarren, Cato et al. 2017). By enabling patient education, support for self-management, motivation, follow-up, feedback and communication, it can prevent, cure or treat many chronic conditions. These features can increase patient motivation and encourage compliance with home exercises and physical activity (Meier, Fitzgerald et al. 2013). Digital behavior change interventions use digital technologies (such as websites, mobile apps, SMS or wearables) to promote and maintain health and have the potential to overcome many barriers compared to in-person programs by providing cost-effective, effective, and accessible information. McCabe et al. 2018). No study has been found in Turkey examining digital interventions or walking programs that include behavior change techniques to increase physical activity in patients with knee osteoarthritis. Considering environmental, cultural and economic factors in this patient group in our society, we think that walking, which we think is the most appropriate physical activity method in terms of cost, accessibility and equipment, should be a permanent behavior. The use of technology to increase physical activity in the era of digitalization is important in terms of addressing the increasing inactivity during the Covid-19 pandemic period. Our aim in the study; To examine the effects of digitally assisted physical activity intervention on pain, functionality and exercise commitment in individuals with knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Knee Osteoarthritis* (ACR criteria)
* 50 years old or over 50 years old
* Pain or discomfort for a total of 28 days or more than 28 days on consecutive or separate days in the past year
* Patients with daily internet access will be included in the study.

Exclusion Criteria:

* Patients with a previous diagnosis of rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis, polymyalgia rheumatica, connective tissue diseases, fibromyalgia or gout
* Patients with a history of using antirheumatic drugs or gout medications
* Patients who have had previous knee arthroplasty and are on the waiting list for total knee or hip replacement surgery
* Patients who have had surgery on the lumbar, hip, knee, foot and ankle joints in the last 12 months
* Patients with a history of acute injury to the knee in the last 6 months
* Patients who have had steroid or hyaluronate injections in the knee in the last 6 months
* Patients with a body mass index of 40 kg/m2 or more
* Patients at risk for unsupervised physical activity

Ages: 50 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Visual analogue scale (VAS) | The pain will be measured at study entry (baseline) after inclusion.
  Pain will be measured using a 10 cm visual analogue scale (VAS). The participants places a mark on the line that best represented their perception of pain at that instant. The VAS score will be measured in cm from the left hand end of the line to the mark.
Visual analogue scale (VAS) | The pain will be measured at the end of intervention (8. week).
  Pain will be measured using a 10 cm visual analogue scale (VAS). The participants places a mark on the line that best represented their perception of pain at that instant. The VAS score will be measured in cm from the left hand end of the line to the mark.
Western Ontario and McMaster Universities Arthritis Index (WOMAC) osteoarthritis index | The WOMAC will be measured at baseline 2 minutes after pain assessment.
  The WOMAC osteoarthritis index is a 24-item scale that examines three dimensions: pain, stiffness, and physical function.
  Each question is scored on a Likert scale as 0=absent, 1=mild, 2=moderate, 3=severe, 4=very severe. The score of each section is calculated on its own and the total score ranges from 0 to 100. High scores indicate increased pain and stiffness and impaired physical function.
Western Ontario and McMaster Universities Arthritis Index (WOMAC) osteoarthritis index | The WOMAC will be measured at the end of intervention (8. week) 2 minutes after pain assessment.
  The WOMAC osteoarthritis index is a 24-item scale that examines three dimensions: pain, stiffness, and physical function.
  Each question is scored on a Likert scale as 0=absent, 1=mild, 2=moderate, 3=severe, 4=very severe. The score of each section is calculated on its own and the total score ranges from 0 to 100. High scores indicate increased pain and stiffness and impaired physical function.
Exercise adherence | Exercise adherence will be measured at the end of intervention (8. week) 2 minutes after WOMAC assessment.
  In the exercise diary, the participant will note the number of steps he takes regularly and the number of exercises he does each day. Patients will be asked to note in their diaries any discomfort they experience in daily life, walking or exercising. The physiotherapist will follow the diaries of the participants included in the walking program assigned to the intervention group each week.

SECONDARY OUTCOMES:
Step count | Step count will be measured at the week before study entry (baseline).
  One week before the intervention, a smart watch will be delivered to the patients and the 1-week step counts will be recorded. Xiaomi Mi Band 3 Smart Wristband will be used for patients to follow their own steps and take notes in their diaries and reach the appropriate number of steps in line with the target given each week.
Step count | Step count will be measured at the 8. week at the end of intervention.
  One week before the intervention, a smart watch will be delivered to the patients and the 1-week step counts will be recorded. Xiaomi Mi Band 3 Smart Wristband will be used for patients to follow their own steps and take notes in their diaries and reach the appropriate number of steps in line with the target given each week.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Akgul H, Birtane M, Tonga E. Effects of a Digitally Supported Physical Activity Intervention in Knee Osteoarthritis: A Pilot Randomized Controlled Trial. Musculoskeletal Care. 2025 Jun;23(2):e70085. doi: 10.1002/msc.70085. PMID 40148223